CLINICAL TRIAL: NCT06489782
Title: Developing a Novel Human Laboratory Paradigm for AUD Medication Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000037693
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model 1 (Experimental): Model 1 examines the impact of alcohol cues and alcohol availability on latency to start drinking and amount consumed of a 0.12 g/dL dose of alcohol during a 2-hour ad-libitum period.
  Interventions: Other: Model 1; Other: Model 2
- Model 2 (Experimental): Model 2 examines the impact of alcohol cues and alcohol availability and a priming dose of alcohol (.04 g/dL) on latency to start drinking and amount consumed of a 0.12 g/dL dose of alcohol during a 2-hour ad-libitum period.
  Interventions: Other: Model 1; Other: Model 2

INTERVENTIONS:
Other: Model 1 — Model 1 examines the impact of alcohol cues and alcohol availability on latency to start drinking and amount consumed of a 0.12 g/dL dose of alcohol during a 2-hour ad-libitum period.
Other: Model 2 — Model 2 examines the impact of alcohol cues and alcohol availability and a priming dose of alcohol (.04 g/dL) on latency to start drinking and amount consumed of a 0.12 g/dL dose of alcohol during a 2-hour ad-libitum period.

SUMMARY:
The intent of the study is to develop two versions of the 'ability to resist' drinking model designed to screen Alcohol Use Disorder (AUD) medications.

DETAILED DESCRIPTION:
Proposed is the development of two versions of the 'ability to resist' drinking model designed to screen AUD medications. Model 1 will examine the impact of alcohol cues and alcohol availability on the 'ability to resist' drinking and subsequent ad-lib drinking. Model 2 (alcohol cues & alcohol availability + low dose prime) on the 'ability to resist' drinking and subsequent ad-lib drinking.

This study will consist of an intake session, a physical exam, and two laboratory sessions. Each laboratory session will start with the presentation of the primes for Model 1 or 2, following which, participants will have the option of initiating an alcohol self-administration session or delaying initiation by five-minute increments for up to 50 minutes in exchange for monetary reinforcement. Subsequently, the alcohol self-administration session entails a 2-hour period in which participants can choose to drink their preferred beverage or receive monetary compensation for alcohol not consumed.

The primary outcome measures for Aim 1 is the latency to start drinking (i.e., ability to resist drinking) and amount consumed during the self-administration sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form;
2. Male or Female Age 21-65;
3. Able to read and write English;
4. Meets DSM-5 criteria for current (past 6 months);
5. Drinking criteria: Males - Drinks > 28 drinks per week and exceeds 4 drinks per day at least once per week; Females -Drinks > 14 drinks per week and exceeds 3 drinks per day at least once per week. Must meet drinking criteria during 30-day period prior to baseline; 6) Laboratory sessions will be scheduled such that participants will not have major responsibilities on the following day which might limit drinking during the self-administration session (e.g., job interview, exam).

Exclusion Criteria:

1. Participants with any significant current medical conditions (neurological, cardiovascular, endocrine, thyroid, renal, liver), seizures, delirium or hallucinations, or other unstable medical conditions including HIV;
2. Current DSM-5 substance use disorder (other than AUD or tobacco use disorder or mild cannabis dependence);
3. A positive test result at intake appointment on urine drug screens conducted for illicit drugs;
4. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD);
5. Suicidal, homicidal or evidence of current (past 6-month) diagnosis of schizophrenia, or bipolar disorder, or psychosis. Participants diagnosed with psychiatric disorders not specifically listed above may be included at the discretion of the study MD as long as the concurrent treatment for the comorbid psychiatric condition does not compromise the study integrity by virtue of its type, duration, or intensity;
6. Only one member per household can participate in the study;
7. Participants likely to exhibit clinically significant alcohol withdrawal during the study. Specifically, we will exclude participants who a) have a history of perceptual distortions, seizures, delirium, or hallucinations upon withdrawal, or b) have a score of > 8 on the Clinical Institute Withdrawal Assessment scale at intake appointments;
8. Individuals who are currently treatment for drinking or who have attempted to quit drinking within the past 3 months in order to exclude participants seeking treatment;
9. Participants who have taken any investigational drug within 4 weeks of intake;
10. Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | 120 minutes
  Means mls of alcohol consumed during 120 minute alcohol self-administration sessions

CONTACTS AND LOCATIONS:
Overall Officials: Sherry McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No